CLINICAL TRIAL: NCT01725529
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Efficacy, Pharmacokinetics, Safety and Tolerability of TMC435 vs. Placebo as Part of a Treatment Regimen Including Peginterferon Alfa-2a and Ribavirin in Treatment-Naïve, Genotype 1 Hepatitis C-Infected Subjects
Brief Title: An Efficacy, Pharmacokinetics, Safety and Tolerability Study of TMC435 as Part of a Treatment Regimen for Hepatitis C-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR017962; TMC435HPC3005 (Other: Janssen R&D Ireland)
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; TMC435; Ribavirin; peginterferon-alpha (PegIFNα-2a)
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Simeprevir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TMC435 150 mg (Experimental): Patients will receive 12 weeks TMC435 150 mg once daily (q.d.) plus peginterferon-alpha (PegIFNα-2a) and ribavirin (RBV), followed by PegIFNα-2a and RBV alone. Response-guided treatment criteria will be used to determine total treatment duration of 24 or 48 weeks for patients in the TMC435 treatment groups. Patients in the control group will continue to receive treatment with PegIFNα-2a and RBV until Week 48.
  Interventions: Drug: TMC435; Drug: Peginterferon-alpha (PegIFNα-2a); Drug: Ribavirin (RBV)
- TMC435 100 mg (Experimental): Patients will receive 12 weeks TMC435 100 mg once daily (q.d.) plus peginterferon-alpha (PegIFNα-2a) and ribavirin (RBV), followed by PegIFNα-2a and RBV alone. Response-guided treatment criteria will be used to determine total treatment duration of 24 or 48 weeks for patients in the TMC435 treatment groups. Patients in the control group will continue PegIFNα-2a and RBV until Week 48.
  Interventions: Drug: TMC435; Drug: Peginterferon-alpha (PegIFNα-2a); Drug: Ribavirin (RBV)
- Control (Placebo Comparator): Patients will receive placebo once daily (q.d.) plus peginterferon-alpha (PegIFNα-2a) and ribavirin (RBV) for 48 weeks.
  Interventions: Drug: Peginterferon-alpha (PegIFNα-2a); Drug: Ribavirin (RBV); Drug: Placebo

INTERVENTIONS:
Drug: TMC435 — TMC435 100 mg or 150 mg capsules taken orally (by mouth) with food once-daily for 12 weeks (Week 12).
  Arms: TMC435 100 mg; TMC435 150 mg
Drug: Peginterferon-alpha (PegIFNα-2a) — PegIFNα-2a (180 micrograms [μg] once weekly) administered as weekly subcutaneous (s.c.) (under the skin) injections of 0.5 mL for 24 or 48 weeks.
Drug: Ribavirin (RBV) — Ribavirin 1000 or 1200 mg/day (taken as 100 mg or 200 mg tablets) depending on body weight (If body weight is < 75 kg the total daily dose of RBV will be 1000 mg, administered as 400 mg intake with food in the morning and 600 mg intake with food in the evening. If body weight is > or = 75 kg the total daily dose will be 1200 mg, administered as 2 x 600 mg per intake with food, morning and evening) for 24 or 48 weeks.
Drug: Placebo — Matching placebo capsules taken orally with food once-daily for 48 weeks.
  Arms: Control

SUMMARY:
The purpose of this study is to provide confirmatory efficacy and safety data of TMC435 as part of a treatment regimen including peginterferon-alpha (PegIFNα-2a) and ribavirin (RBV) in patients with genotype 1 Hepatitis C virus (HCV) infection.

DETAILED DESCRIPTION:
This is a multicenter, randomized (study drug is assigned by chance), double-blind (neither sponsor, physician nor patient knows the name of the assigned study drug), Phase III study to compare the efficacy, tolerability and safety of TMC435 (in development for treatment of chronic hepatitis C virus [HCV] infection) versus placebo (a preparation containing no drug used as control) as part of a treatment regimen including peginterferon-alpha (PegIFNα-2a) and ribavirin (RBV) (both current therapies for HCV) in adult treatment-naïve patients (patients who have never taken HCV medications) with genotype 1 Hepatitis C virus (HCV) infection. The study will consist of a screening period with a maximum duration of 6 weeks, a response guided 24- or 48-week (TMC435 treatment groups) or 48-week (control group) treatment period, and a post-therapy follow-up period up to 72 weeks after the start of treatment. Patients will be randomly assigned in a 1:1:1 fashion to receive TMC435 or placebo, stratified by HCV genotype 1 subtype and IL28B genotype within each country. In the first 24 weeks, patients will receive 12 weeks TMC435 100 or 150 mg or placebo once-daily (q.d.) plus PegIFNα-2a plus RBV, after which they will continue with PegIFNα-2a and RBV. Response-guided treatment criteria will be used to determine PegIFNα-2a and RBV total treatment duration of 24 or 48 weeks for patients in the TMC435 treatment groups. In the control group, all patients will be required to complete 48 weeks of treatment with PegIFNα-2a and RBV. In all 3 treatment groups, there will be a post-therapy follow-up period up to 72 weeks after the start of treatment. The total study duration for each patient will be a maximum of 78 weeks (including the 6-week screening period).

ELIGIBILITY:
Inclusion Criteria:

* A liver biopsy within 3 years prior to the screening visit (or between screening and day of randomization) with histology consistent with chronic Hepatitis C virus (HCV) infection
* Presence of contraindications for a liver biopsy in patients who are otherwise deemed eligible for participation does not exclude the patient from participation
* Genotype 1 HCV infection (confirmed at screening)
* Plasma HCV RNA of > 10,000 IU/mL at screening

Exclusion Criteria:

* Prior treatment with any approved or investigational drug for the treatment of hepatitis C
* Co-infection with hepatitis B virus or human immunodeficiency virus (HIV)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2012-11; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (21):
- China (16):
  - Beijing
  - Changchun
  - Changsha
  - Chengdu
  - Chongqing
  - Guangzhou
  - Hangzhou
  - Harbin
  - Jinan
  - Lanzhou
  - Nanjing
  - Shanghai
  - Shenyang
  - Tianjin
  - Wuhan
  - Zhengzhou
- South Korea (5):
  - Busan
  - Chuncheon, Gangwon-Do
  - Gyeongsangnam-Do
  - Incheon
  - Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matching to TMC435 100 milligram (mg) and TMC435 150 mg for 12 weeks once daily (q.d.) plus peginterferon-alpha (PegIFNa-2a) and ribavirin (RBV) for 48 weeks.
- Simeprevir (TMC435) 100mg: Participants received TMC435 100 mg once daily (q.d.) for 12 weeks plus peginterferon-alpha (PegIFNα-2a), ribavirin (RBV) and Placebo matching to TMC435 150 mg, followed by PegIFNα-2a and RBV alone. Response-guided treatment criterion was used to determine total treatment duration of 24 or 48 weeks for participants in the TMC435 treatment groups.
- Simeprevir (TMC435) 150mg: Participants received TMC435 150 mg once daily (q.d.) for 12 weeks plus peginterferon-alpha (PegIFNα-2a), ribavirin (RBV) and Placebo matching to TMC435 100 mg, followed by PegIFNα-2a and RBV alone. Response-guided treatment criterion was used to determine total treatment duration of 24 or 48 weeks for participants in the TMC435 treatment groups.
Period: Overall Study
Arm/Group | Placebo | Simeprevir (TMC435) 100mg | Simeprevir (TMC435) 150mg
Started | 152 | 153 | 152
Completed | 137 | 137 | 142
Not Completed | 15 | 16 | 10
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 12 | 14 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Simeprevir (TMC435) 100mg | Simeprevir (TMC435) 150mg | Total
Number analyzed (Participants) | 152 | 153 | 152 | 457
Age, Continuous [Median (Full Range); unit: years] | 45 [18 to 68] | 45 [18 to 68] | 44 [19 to 68] | 45 [18 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 67 | 75 | 221
  Male | 73 | 86 | 77 | 236

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After End of Study Drug Treatment (SVR12)
Description: Participants considered to have achieved SVR12 if both conditions are met: 1). the hepatitis C virus ribonucleic acid (HCV RNA) is less than (<) lower limit of quantification (LLOQ; 25 international unit per milliliter [IU/mL]) undetectable at end of treatment and, 2). the HCV RNA is < LLOQ detectable or undetectable at 12 weeks after the planned end of study drug treatment.
Time Frame: 12 weeks after the end of treatment (EOT: Week 24 or 48)
Population: Intent-to-treat (ITT) population included all the randomized participants who took at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Simeprevir (TMC435) 100mg | Simeprevir (TMC435) 150mg
Number analyzed (Participants) | 152 | 153 | 152
Percentage of participants | 75.7 | 88.9 | 90.8

2. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks After End of Study Drug Treatment (SVR24)
Description: Participants considered to have achieved SVR24 if both conditions are met: 1). the hepatitis C virus ribonucleic acid (HCV RNA) is less than (<) lower limit of quantification (LLOQ;25 IU/mL) undetectable at end of treatment and, 2). the HCV RNA is < LLOQ detectable or undetectable at 24 weeks after the planned end of study drug treatment.
Time Frame: 24 weeks after the end of treatment (EOT: Week 24 or 48)
Population: ITT population included all the randomized participants who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Simeprevir (TMC435) 100mg | Simeprevir (TMC435) 150mg
Number analyzed (Participants) | 152 | 153 | 152
percentage of participants | 75.0 | 88.9 | 90.8

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at Week 72 (SVRW72)
Time Frame: Week 72
Population: ITT population included all the randomized participants who took at least 1 dose of study drug. 'N' (number of participants analyzed) signifies those participants who were analyzed for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Simeprevir (TMC435) 100mg | Simeprevir (TMC435) 150mg
Number analyzed (Participants) | 152 | 153 | 152
percentage of participants | 75.0 | 87.6 | 90.1

4. Secondary Outcome: Percentage of Participants With On-treatment Failure
Description: A participant with on-treatment failure refers to a participant with confirmed detectable HCV RNA at the end of treatment.
Time Frame: End of Treatment (EOT: Week 24 or 48)
Population: ITT population included all the randomized participants who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Simeprevir (TMC435) 100mg | Simeprevir (TMC435) 150mg
Number analyzed (Participants) | 152 | 153 | 152
percentage of participants | 12.5 | 3.3 | 3.3

5. Secondary Outcome: Percentage of Participants With Viral Breakthrough
Description: The number of patients who experience viral breakthrough will be determined by measuring Hepatitis C virus (HCV) ribonucleic acid (RNA) levels in plasma. Viral breakthrough was defined as a confirmed increase of >1 log10 IU/mL in HCV RNA level from the lowest level reached, or a confirmed HCV RNA level of >100 IU/mL in subjects whose HCV RNA levels had previously been below the limit of quantification (<25 IU/mL detectable) or undetectable (<25 IU/mL undetectable) while on study treatment.
Time Frame: Week 24 or 48 (End of Treatment)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Simeprevir (TMC435) 100mg | Simeprevir (TMC435) 150mg
Number analyzed (Participants) | 152 | 153 | 151
percentage of participants | 2.0 | 2.6 | 2.6

6. Secondary Outcome: Percentage of Participants With Viral Relapse
Description: Viral relapse was defined as undetectable HCV RNA at the actual end of treatment and last HCV RNA measurement during follow-up ≥25 IU/mL.
Time Frame: 72 weeks after the EOT (Week 24 or 48)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Simeprevir (TMC435) 100mg | Simeprevir (TMC435) 150mg
Number analyzed (Participants) | 131 | 142 | 141
percentage of participants | 11.5 | 1.4 | 2.8

7. Secondary Outcome: Percentage of Participants With On-treatment Normalization of Alanine Aminotransferase Level
Description: Percentage of participants with on-treatment normalization of alanine aminotransferase level were assessed.
Time Frame: 72 weeks after the EOT (Week 24 or 48)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Simeprevir (TMC435) 100mg | Simeprevir (TMC435) 150mg
Number analyzed (Participants) | 91 | 79 | 89
percentage of participants | 85.7 | 86.1 | 89.9

ADVERSE EVENTS:
Time Frame: up to 4 weeks after End of treatment (EOT: Week 24 or Week 48)
Arm/Group | Placebo | Simeprevir (TMC435) 100mg | Simeprevir (TMC435) 150mg
Serious Adverse Events (participants affected / at risk) | 9/152 | 5/153 | 5/152
Other Adverse Events (participants affected / at risk) | 149/152 | 149/153 | 149/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=152) | Simeprevir (TMC435) 100mg (N=153) | Simeprevir (TMC435) 150mg (N=152)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cholesterosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Incision site infection (Infections and infestations) | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0
Chronic hepatitis C (Infections and infestations) | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Undifferentiated connective tissue disease (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=152) | Simeprevir (TMC435) 100mg (N=153) | Simeprevir (TMC435) 150mg (N=152)
Neutrophil count decreased (Investigations) | 94 | 87 | 84
White blood cell count decreased (Investigations) | 81 | 77 | 80
Platelet count decreased (Investigations) | 63 | 57 | 73
Haemoglobin decreased (Investigations) | 57 | 46 | 47
Blood bilirubin increased (Investigations) | 27 | 31 | 54
Bilirubin conjugated increased (Investigations) | 5 | 10 | 33
Red blood cell count decreased (Investigations) | 25 | 23 | 20
Lymphocyte count decreased (Investigations) | 20 | 19 | 18
Haematocrit decreased (Investigations) | 19 | 17 | 17
Alanine aminotransferase increased (Investigations) | 27 | 14 | 19
Blood bilirubin unconjugated increased (Investigations) | 8 | 11 | 21
Aspartate aminotransferase increased (Investigations) | 24 | 12 | 15
Monocyte count decreased (Investigations) | 11 | 12 | 13
Blood calcium decreased (Investigations) | 9 | 9 | 9
Neutrophil percentage decreased (Investigations) | 5 | 10 | 8
Low density lipoprotein decreased (Investigations) | 5 | 6 | 11
Mean cell haemoglobin concentration decreased (Investigations) | 9 | 9 | 8
Mean cell volume increased (Investigations) | 9 | 10 | 7
Blood cholesterol decreased (Investigations) | 6 | 6 | 9
Blood lactate dehydrogenase increased (Investigations) | 10 | 4 | 6
Gamma-glutamyltransferase increased (Investigations) | 14 | 2 | 3
Blood potassium decreased (Investigations) | 8 | 1 | 3
Pyrexia (General disorders) | 46 | 29 | 38
Fatigue (General disorders) | 36 | 35 | 28
Influenza like illness (General disorders) | 19 | 20 | 19
Asthenia (General disorders) | 7 | 8 | 7
Anaemia (Blood and lymphatic system disorders) | 53 | 38 | 44
Neutropenia (Blood and lymphatic system disorders) | 32 | 28 | 31
Thrombocytopenia (Blood and lymphatic system disorders) | 22 | 20 | 15
Leukopenia (Blood and lymphatic system disorders) | 16 | 13 | 16
Rash (Skin and subcutaneous tissue disorders) | 27 | 27 | 30
Alopecia (Skin and subcutaneous tissue disorders) | 26 | 21 | 26
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 23 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 22 | 21 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 8 | 5
Headache (Nervous system disorders) | 28 | 23 | 16
Nausea (Gastrointestinal disorders) | 10 | 8 | 8
Diarrhoea (Gastrointestinal disorders) | 7 | 4 | 10
Abdominal pain upper (Gastrointestinal disorders) | 10 | 4 | 9
Decreased appetite (Metabolism and nutrition disorders) | 16 | 17 | 11
Hyperbilirubinaemia (Hepatobiliary disorders) | 4 | 14 | 10
Upper respiratory tract infection (Infections and infestations) | 12 | 4 | 13
Nasopharyngitis (Infections and infestations) | 10 | 2 | 5
Insomnia (Psychiatric disorders) | 18 | 8 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 8 | 8
Hypothyroidism (Endocrine disorders) | 9 | 3 | 6
Vertigo (Ear and labyrinth disorders) | 10 | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.